CLINICAL TRIAL: NCT05646810
Title: Impact of Peripheral Afferent Input on Central Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 39451
Record Dates: First submitted 2022-11-14; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-11

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases; Syringomyelia
Keywords: central pain; peripheral afferent input; neuropathic pain; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Syringomyelia; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): Nerve block
  Interventions: Diagnostic Test: Lidocaine (10 mg/ml)
- Isotonic saline (Placebo Comparator): Nerve block
  Interventions: Diagnostic Test: Isotonic saline

INTERVENTIONS:
Diagnostic Test: Lidocaine (10 mg/ml) — Lidocaine (10 mg/ml) will be injected according to established protocols using ultrasound guidance and an aseptic technique by an experienced anesthesiologist.
  Arms: Lidocaine
Diagnostic Test: Isotonic saline — Isotonic saline will be injected according to established protocols using ultrasound guidance and an aseptic technique by an experienced anesthesiologist.
  Arms: Isotonic saline

SUMMARY:
The overarching aim of this study is to investigate the contribution of peripheral afferent input to spontaneous and evoked central neuropathic pain after a spinal cord lesion or disease.

DETAILED DESCRIPTION:
A key question that has been subject to longstanding debates in the field relates to the sites and mechanisms within the peripheral or central nervous system that potentially perpetuate chronic spontaneous and evoked central neuropathic pain. The investigators hypothesize that spontaneous central neuropathic pain depends on continuous, "physiological" somatosensory input from the painful body region in the periphery. Thus, spontaneous central neuropathic pain results from pathological gain control in central somatosensory networks with decreased activation thresholds for thermo- and mechanosensitive peripheral afferents.

ELIGIBILITY:
Inclusion Criteria:

* Definite central neuropathic pain according to current diagnostic algorithms involving at least both feet or both hands bilaterally and symmetrically with regard to the expected neuroanatomical distribution of the nerve block.
* Patients with spinal cord injury. For patients with pain in both legs, the injury has to be incomplete. For patients with pain in both arms, the injury can be complete or incomplete. The pain in the area that will be investigated (region of interest) has to be in an area with at least some preservation of sensation
* An intensity of spontaneous pain of ≥4 NRS [0-10] in the region of interest during the screening visit and at the day of the intervention.
* Participant is able and willing to give informed consent.
* For female subjects of childbearing potential: A negative pregnancy test and either use of highly effective contraception or sexual abstinence

Exclusion Criteria:

* Conus/cauda involvement or evidence of peripheral neuropathic pain due to documented peripheral lesion.
* Other known neurological and psychiatric conditions
* History or symptoms of significant diseases that may confound the measurements or represent contra-indications for the intervention (e.g., neuropathy following cancer or metabolic diseases such as diabetes mellitus, liver diseases, and kidney diseases.
* Cardiovascular diseases that preclude the anaesthetic intervention (e.g., arrythmias).
* Concomitant nociceptive pain within the innervation territory of the planned nerve block.
* Unable to understand and speak Danish
* Changes in pain medication within the last 4 weeks prior to the intervention.
* Treatment with warfarin or other blood thinning medications, that contraindicates regional anesthesia if the treating physician cannot recommend that such treatments are paused for at least 7 days before the study day
* Infection or skin disease in planned injection area
* Allergy for local anesthetics
* Pregnancy or lactation.
* Alcohol or drug abuse
* Pain intensity below 4 in the region of interest at the baseline measurement before the nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Indication of most pain relief | 40 minutes
  Limb with most pain relief on Numerical Rating Scale (NRS) [0-10, 0=no pain 10=worst pain imaginable] 40 minutes after nerve block

SECONDARY OUTCOMES:
Intensity on Numerical Rating Scale (NRS) [0-10, 0=no pain 10=worst pain imaginable] of spontaneous pain | 90 minutes
  Intensity on Numerical Rating Scale (NRS) [0-10, 0=no pain 10=worst pain imaginable] of spontaneous pain in the pre-specified region covered by the block 40, 60 and 90 min after the nerve block compared to baseline
Pain relief 45 min after the nerve block | 45 minutes
  Pain relief 45 min after the nerve block using a 6-point verbal scale ranging from worse pain to no, little, moderate, good and complete pain relief (-1 to 4)
Pain extent [% of body surface on standardized pain drawings] 50 minutes after the nerve block | 50 minutes
  Pain extent will be mapped on standardized pain drawings 50 minutes after the nerve block compared to baseline
Pain descriptors 50 minutes after the nerve block | 50 minutes
  Pain descriptors (burning, squeezing, pins and needles, tingling, stabbing, electrical shocks) are captured 50 minutes after the nerve block compared to baseline
Area [% of pain extent] of hypersensitivity to thermal and nociceptive stimuli | 95 minutes
  Area of hypersensitivity [% of pain extent] to warm (40°C) and cold (20°C) thermo rollers (Somedic AB, Hörby, Sweden), pinprick (Semmes-Weinstein monofilament no 5.88 (bending force 75.9 g/745 mN)), and brush (SENSELab Brush-05; Somedic AB, Hörby, Sweden), if any, 55 and 95 min after nerve block compared to baseline
Intensity of hypersensitivity on Numerical Rating Scale (NRS) [0-10, 0=no pain 10=worst pain imaginable] to thermal and nociceptive stimuli | 95 minutes
  Intensity of hypersensitivity on Numerical Rating Scale (NRS) [0-10, 0=no pain 10=worst pain imaginable] to warm (40°C) and cold (20°C) thermo rollers (Somedic AB, Hörby, Sweden), pinprick (Semmes-Weinstein monofilament no 5.88 (bending force 75.9 g/745 mN)), and brush (SENSELab Brush-05; Somedic AB, Hörby, Sweden), if any, 55 and 95 min after nerve block compared to baseline

OTHER OUTCOMES:
Plasma lidocaine concentrations | 40 minutes
  Plasma lidocaine concentrations approx. 40 min after the block.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Rosner, MD, Principal Investigator — Danish Pain Research Center, Department of Clinical Medicine, Aarhus University

IPD SHARING:
Plan to Share IPD: No